CLINICAL TRIAL: NCT04240509
Title: Defining the PrEP Care Continuum Among Recently Incarcerated Men at High-Risk for HIV Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrEP Care-Gilead
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir — Incarcerated men identified at high risk for HIV transmission will be given a 30-day supply of the study drug and will be provided with patient navigation to follow up care upon release.

SUMMARY:
Background: Several major studies have demonstrated the success of Truvada as pre-exposure prophylaxis (PrEP) in preventing HIV infection.The CDC guidelines recommend PrEP for people who are at elevated risk of HIV including men who have sex with men (MSM) and people who use injection drugs. People who are incarcerated bear a disproportionate of disease burden, including HIV. Furthermore, men who have been involved with the criminal justice system are more likely to engage in risky behaviors following their release, including condomless sex with partners of unknown serostatus, and injection drug use.

The incarceration setting provides a place to engage men who may be at risk of HIV after they are released.

Following release, community clinics, including the STD clinic at The Miriam Hospital (TMH) Immunology Center, that perform routine testing for HIV and other sexually transmitted diseases (STDs) may be ideal settings to engage vulnerable populations in care, including PrEP.

Despite the demonstrated clinical efficacy of PrEP in reducing HIV transmissions, few clinical programs have piloted the use of PrEP in real-world settings, particularly criminal justice settings. Furthermore, studies demonstrate numerous challenges to PrEP uptake and adherence, including a lack of access or discontinuing care. Engaging at risk men in PrEP care before they leave prison and potentially lost to care during the transition may increase uptake, adherence, and retention.

Objective: This study protocol will evaluate a clinical program that aims to prevent new HIV infections among recently-incarcerated men using a once daily dosing of tenofovir/emtricitabine (Truvada) as pre-exposure prophylaxis (PrEP). This protocol presents an overview of the clinical program, which uses standard-of-care clinical practices and Centers for Disease Control and Prevention (CDC) guidelines for prescribing and monitoring PrEP.

Male inmates at the Rhode Island Department of Corrections (RIDOC) will be screened for HIV risk and, if eligible and interested, will be prescribed and given a one-month supply of PrEP shortly before their release, and receive follow up care at The Miriam Hospital (TMH) Immunology Center following their release.

ELIGIBILITY:
Inclusion Criteria:

* Current men committed at the RIDOC (aged 18 and above); HIV negative; meet CDC indications for PrEP use (based on risk criteria before they were sentenced); interested in taking PrEP; and are able to voluntarily consent to be treated will be included

Exclusion Criteria:

* Individuals who are younger than 18 years old; are HIV positive, Hepatitis B Virus positive or have a CrCl<60; or unable to provide voluntary consent will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number retained in PrEP care | 6 months
  The primary outcome of the proposed study will be the number of individuals retained in PrEP care at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States